

IVFarma LLC Nauchny proezd, 20, 2 117246 Moscow Russia Tel/fax +7(499)645-53-42 OGRN: 1127746597527 INN: 7728815153

| Official Title of the study: | An Observational Study "FOLLITROPIN" Comparing the Efficacy of Follitropin Alpha Biosimilar: The Realworld Data |
|---|---|
| Ethics approval and consent to participate: | Women with established causes of infertility and indications for the use of ART methods, according to the Order of the Ministry of Health of the Russian Federation "On the use of assisted reproductive technologies, contraindications and limitations to their use" No. 107 n dated August 30, 2012. |
| Unique Protocol ID: | IVF-2020 |
| NCT number: | ClinicalTrials.gov Identifier: NCT04854707 Date of registration: April 22, 2021, retrospectively registered. |
| General Manager/IVFarma LLC<br>Mikhail Polzikov (PhD) | Study protectol approval: 10.01.2021 |

## STUDY SUMMARY

| Study title: | An Observational Study "FOLLITROPIN" Comparing the Efficacy of Follitropin Alpha Biosimilar: The Real-world Data |
|---|---|
| Study type: | Phase IV |
| Test product | TN: Primapur® INN: follitropin alpha Dosage form: solution for subcutaneous injection Pharmaceutical form: pre-filled disposable syringe containing follitropin alpha 66 μg (900 IU), 33 μg (450 IU), 22 μg (300 IU), Manufacturer: Zavod Medsintez LLC, Russia |
| Ethical and legal aspects: | <ul> <li>This study conducted in strict accordance with the following international and Russian documents:</li> <li>1. Principles of the World Medical Association Declaration of Helsinki (Fortaleza, Brazil, 2013).</li> <li>2. Constitution of the Russian Federation.</li> <li>3. Federal Law "On the fundamentals of protecting the health of citizens in the Russian Federation" dated November 21, 2011 No. 323-FZ, 2011.</li> <li>4. Federal Law "On the Circulation of Medicines" No. 61-FZ dated 12 April 2010.</li> <li>5. Federal Law "On personal data" No. 152-FZ dated July 27, 2006.</li> <li>6. Order of the Ministry of Health of the Russian Federation "On the use of assisted reproductive technologies, contraindications and limitations to their use" No. 107 n dated August 30, 2012.</li> </ul> |
| Study goals: | To investigate the efficacy of follitropin alpha biosimilar therapy (Primapur®) in nonselected real-world population. |
| Study objectives: | The efficacy and safety of biosimilar follitropin alpha have been demonstrated in randomized blinded prospective clinical trials of phases I and III. Unfortunately, there is a gap between the clinical trials and real clinical practice data. The real-world patient data helps to create an evidence-based background for successful implementation of medicine at everyday practice in a nonselected population. The ovarian stimulation (OS) protocols included: monotherapy protocols with using only follitropin alpha biosimilar (Primapur®); mixed protocols (recombinant and urinary-derived gonadotropins) and follitropin alpha biosimilar; short protocols with using antagonists of gonadotropin-releasing hormone (GnRH) and long protocols with |

| | GnRH agonists. The stimulation protocols were analyzed |
|---|---|
| | with Primapur® application for at least 5 days. |
| Study design: | Retrospective, observational (non-interventional), anonymized, |
| | cohort study |
| Number of patients | 5500 patients |
| realiser of patients | 3300 patients |
| Study centers | 35 in vitro fertilization (IVF) clinics in the Russian Federation |
| Study population: | Women aged 20-43 with established causes of infertility and indications |
| | for the use of assisted reproductive technologies (ART) and ovarian |
| | stimulation. |
| Inclusion criteria: | 1. Women with established causes of infertility and indications for the |
| | use of ART methods, according to the Order of the Ministry of Health |
| | of the Russian Federation "On the use of assisted reproductive |
| | technologies, contraindications and limitations to their use" No. 107 n |
| | dated August 30, 2012. |
| | 2. Infertility due to female and/or male factor. |
| | 3. Presence of ovaries accessible for aspiration of follicles. |
| | 4. Anatomical and functional capability of uterus to bear pregnancy. |
| Exclusion criteria: | <ol> <li>Women with established contraindications to the use of ART methods, according to the Order of the Ministry of Health of the Russian Federation "On the use of assisted reproductive technologies, contraindications and limitations to their use" No. 107 n dated August 30, 2012.</li> <li>Presence of pregnancy</li> <li>Hypersensitivity to follitropin alpha and other gonadotropins or excipients.</li> <li>Ovarian cysts (not associated with polycystic ovarian syndrome), uterine hemorrhage of unclear etiology</li> <li>Premature ovarian failure</li> <li>Presence of clinically significant systemic disease</li> <li>Presence of chronic cardiovascular, hepatic, renal or pulmonary disease</li> <li>Neoplasia</li> <li>Narcomania, alcoholism</li> </ol> |
| Dosage and duration of | Drug: Follicle Stimulating Hormone/Luteinizing Hormone |
| treatment; route of | Overall ovarian stimulation protocols with follitropin alpha |
| administration: | biosimilar for at least 5 days (100-300 IU) and other recombinant |
| | follitropins and menotropins, short (antagonists of GnRH) or long |
| | protocols (agonist of GnRH). |
| Concomitant therapy: | All patients received approved medication by physician, accordingly |
| | to National guidelines. |

## Efficacy evaluation criteria: **Study endpoints per patient: Primary point:** Total number of aspirated oocytes. Incidence of clinical pregnancies (up to 6 weeks after the embryo(s) transfer). **Secondary points:** Number of mature oocytes (MII stage). Number of fertilized oocytes (zygotes with 2PN). Total dose of a follitropin alpha biosimilar injected (IU). of serious adverse events e.g., Safety evaluation criteria: Incidence ovarian hyperstimulation syndrome (%) with hospitalization. Incidence of the adverse event, such as injection site pain (%). 1. Monoprotocols: follitropin alpha biosimilar only **Groups/arms to compare:** antagonists/agonists of GnRH (The ovarian stimulation (OS) protocols included monotherapy protocols with using follitropin alpha biosimilar only and antagonists/agonists of of gonadotropin-releasing hormone (GnRH): ganirelix, cetrorelix, triptorelin, buserelin). 2. Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH. (The OS protocols included: mixed protocols (recombinant with addition of urinary-derived gonadotropins) and antagonists/agonists of GnRH (ganirelix, cetrorelix, triptorelin, buserelin), where follitropin alpha biosimilar used for at least 5 days during OS). 3. Monoprotocols: follitropin alpha biosimilar only and antagonists of GnRH (The OS protocols included: monotherapy protocols with using only follitropin alpha biosimilar and antagonists of GnRH). 4. Monoprotocols: follitropin alpha biosimilar only and agonist of GnRH (The OS protocol included: monotherapy protocols with using only follitropin alpha biosimilar and agonists of GnRH). 5. The overall protocols (The OS protocols included: (1) Monoprotocols: follitropin alpha biosimilar only and antagonists/agonists of GnRH, (2) Mixed protocols: recombinant and urinary-derived gonadotropins and antagonists/agonists of GnRH).



In order to compare two groups of normally distributed quantitative data, the Student's t-test will be used; if quantitative data distribution differs from normal values, the Mann-Whitney U test will be used. For intergroup comparisons by qualitative characteristics, the Fisher's exact test will be used.

## Applicable significance level

In this study, the indicators are considered statistically significant at the bilateral p-value level <0.05.